CLINICAL TRIAL: NCT03015597
Title: Addition of Contingency Management to Stop Smoking Services for Patients Undergoing Treatment for Opiate Addiction: a Randomised Controlled Pilot Study
Brief Title: Pilot Study of Contingency Management for Smoking Cessation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 171709
Record Dates: First submitted 2016-09-28; First posted 2017-01-10 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2016-12

CONDITIONS: Smoking; Tobacco Smoking; Smoking, Tobacco; Smoking Cessation; Opiate Addiction; Opiate Dependence
Keywords: Smoking; Tobacco Smoking; Smoking, Tobacco; Smoking Cessation; Opiate Addiction; Opiate Dependence; Contingency Management
MeSH Terms: conditions — Smoking; Tobacco Smoking; Smoking Cessation; Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contingency Management: smoking (Experimental): Contingency Management: smoking
  Participants receive rewards contingent on biochemical verification of tobacco smoking abstinence
  Interventions: Behavioral: Contingency Management
- Contingency Management: attendance (Placebo Comparator): Contingency Management: attendance
  Participants receive rewards contingent on attending the stop smoking clinic (independent of smoking status)
  Interventions: Behavioral: Contingency Management

INTERVENTIONS:
Behavioral: Contingency Management — Contingency management is a behavioural intervention based on the principals of operant conditioning that is widely used in the addictions field. At the most basic level, contingency management works by providing rewards as reinforcement for desired behaviours. In the current study, the desired behaviours are either attendance at the clinic and abstinence from tobacco smoking, or just attendance at the clinic, dependent on the arm of the trial that participants are randomised to. Participants in the experimental condition will receive shopping vouchers for attending the clinic and providing a breath CO recording of <10ppm. Participants in the control condition will receive shopping vouchers for attending the clinic, regardless of their breath CO recording results.

SUMMARY:
The purpose of this study is to see whether contingency management (CM) can be successfully added as an adjunct treatment to standard stop smoking services in outpatients undergoing treatment for opiate addiction. Forty tobacco smoking patients undergoing treatment for opiate addiction will be stratified to a CM intervention for either smoking abstinence or attendance at the clinic, whilst also receiving usual stop smoking services cessation treatment. The intervention will run for five weeks and participants will be followed up six months after the beginning of the study.

DETAILED DESCRIPTION:
The study aims to investigate whether a contingency management (CM) intervention can be added to usual NHS stop smoking services (SSS) treatment, in patients undergoing treatment for opiate addiction.

The SSS at the treatment centre follows the standard treatment program set out by the National Centre for Smoking Cessation and Training (NCSCT) and the NICE guidelines for smoking cessation. Service users taking part in the SSS attend one meeting per week for six weeks. In the first meeting with a cessation worker the client completes baseline information about the client's age, gender, ethnicity, employment, motivation to quit, past quit attempts and current smoking behaviour), and sets a quit date for the following week. For the remaining four weeks clients attend the clinic to receive behavioural support. Nicotine replacement therapy (NRT) is available free of charge to all individuals engaged with SSS. During the six weeks of treatment, service users are given a week's supply of NRT at a time. At the end of the six weeks, service users are given a two week supply of NRT before exiting the SSS treatment. NRT use is recorded throughout SSS treatment. Clients' breath carbon monoxide (CO) levels are also measured at the initial visit and at each subsequent visit over the next 5 weeks in order to biochemically verify self-reported abstinence from smoking (CO<10ppm).

The CM intervention that this study will run as an adjunct to the SSS,. The 40 participants will be randomised into either experimental (CM for abstinence) or control (CM for attendance) conditions at intake. Randomisation will be stratified based on participants' current smoking frequency (between 10 and 20 per day, and more than 20 per day). The intervention will run for five weeks in total, with randomisation occurring at visit 1, and the intervention beginning in week two of the SSS treatment and ending in week six. Participants will be rewarded for smoking abstinence in the experimental condition, and for attending the SSS clinic in the control condition. For the experimental condition smoking abstinence will be defined as a breath CO reading of <10ppm, and for the control condition attendance will be defined as attending the SSS clinic once a week. Rewards will be administered by a researcher to ensure cessation workers are not aware of group allocation.

The intervention will employ an 'escalating with reset' schedule, Reward values will be the same in both conditions. In escalating with reset CM, rewards escalate in a set increment value for each successive verified display of the desired behaviour. When the desired behaviour is not observed, no reward is given, and the reward value for the next verified display of the desired behaviour is reset to that of the initial reward. Reward values then begin to rise again in the same way as before.

Six months after their set quit date, participants will be contacted by the PI to ascertain their self-reported smoking status. In order to test the optimal follow up method, participants will be pseudo-randomised to be contacted by text and phone call, or email and phone call. All participants will also be asked to return to the clinic in order to have their breath CO levels tested to verify this. Once this is done, participants will have completed their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Want to quit smoking
* Between 18 and 65 years old
* Undergoing current pharmacological treatment for opiate addiction
* Smoke a minimum of 10 cigarettes per day
* Provide informed consent.

Exclusion Criteria:

* Insufficient English skills to understand study protocols
* Currently undergoing treatment for drugs other that opiates or tobacco
* Taking part in other research

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-10; Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of participants completing treatment in each condition | 6 weeks
  Number of participants completing treatment in each condition

SECONDARY OUTCOMES:
Percentage of negative samples | Each week throughout intervention (weeks 1-6) and at 6 month follow up
  Percentage of biochemically verified (exhaled air carbon monoxide) negative breath samples b) Biochemically verified (exhaled air carbon monoxide) point prevalence smoking abstinence
Longest duration of abstinence | Each week throughout intervention (weeks 1-6) and at 6 month follow up
  Number of consecutively biochemically verified (exhaled air carbon monoxide) negative breath samples
Point Prevalence abstinence | Each week throughout intervention (weeks 1-6) and at 6 month follow up
  Biochemically verified (exhaled air carbon monoxide) point prevalence smoking abstinence

CONTACTS AND LOCATIONS:
Overall Officials: Ann McNeill, PhD, Study Director — King's College London
Locations (1):
- Lorraine Hewitt Hosue, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Permission is not being sought for this from participants to expedite recruitment

REFERENCES:
- [Derived] Ainscough TS, Brose LS, Strang J, McNeill A. Contingency management for tobacco smoking during opioid addiction treatment: Implementation challenges. Drug Alcohol Rev. 2021 May;40(4):658-661. doi: 10.1111/dar.13216. Epub 2020 Nov 24. PMID 33233020